CLINICAL TRIAL: NCT03150134
Title: Early Tapering of Immunosuppressive Agents After Allogeneic Hematopoietic Stem Cell Transplantation Can Improve the Survival of Patients With Advanced Acute Myeloid Leukemia.
Brief Title: Early Tapering of Immunosuppressive Agents to Immunomodulation to Improve Survival of AML Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Yang Jun, Principal Investigator, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017KY21
Record Dates: First submitted 2017-05-05; First posted 2017-05-12 (Actual); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Acute Myeloid Leukemia; Disorder Related to Bone Marrow Transplantation
Keywords: Acute Myeloid Leukemia; transplantation; allogeneic transplantation; immunosuppressive agents
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Cyclosporine; Immunosuppressive Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- early reduction (Experimental): Usually in the absence of GvHD, immunosuppressive drugs(Cyclosporine) were gradually reduced by 6 weeks and discontinued in three months after transplant in the advanced patients while immunosuppressive agents were gradually reduced by 2 months and discontinued in four months after transplant in the advanced patients in haploidentical SCT even if complete donor chimerism (CDC) achieved. If donor chimerism had not achieved CDC with no significant acute GVHD at four weeks after HSCT, immunosuppressive agents were gradually reduced. If GvHD was present during the time of immunosuppressive agents reduction, CsA was added again and tapering was done over longer periods.
  Interventions: Drug: Cyclosporine
- routine reduction (Placebo Comparator): Arm/Group Descriptions.Immunosuppressive drugs(cyclosporine) were routine reduced by 3 months and discontinued in the 5 months without GvHD in the CR group. We used the result of chimerism as the reference.
  Interventions: Drug: routine reduction of immunosuppressive drugs(cyclosporine)

INTERVENTIONS:
Drug: Cyclosporine — Patients with advanced AML received early tapering of immunosuppressive drugs(Cyclosporine)
  Other Names: immunosuppressive agents
  Arms: early reduction
Drug: routine reduction of immunosuppressive drugs(cyclosporine) — patients with AML in CR were given the routine reduction of immunosuppressive drugs(cyclosporine)
  Other Names: cyclosporine
  Arms: routine reduction

SUMMARY:
Early reduction of immunosuppressive agents after HLA matched donor transplantation can improve the survival of advanced stage acute myeloid leukemia.

single-center, open clinical study

DETAILED DESCRIPTION:
Although 60-80% of AML patients can achieve complete remission through conventional chemotherapy, relapse is still a common problem. For patients unlikely to respond, re-induction attempts may be dismal, leading to more organ toxicity and increased tumor resistance. In addition, 10% to 40% of patients are primary induction failure (PIF) or resistant disease. AML with PIF or relapse still represents one of the most poor outcomes. In such settings, allogeneic transplantation(allo-HSCT) remains the best prospect of curative potential in a small percentage of patients.

However, several retrospective studies have reported long-term survival rates only of 10% to 40% for patients with AML not in remission at the time of allo-HSCT. Michel Duval et al reported that leukemia progression was the single most frequent cause of failure( 42% for AML) for these patients with advanced disease. It is widely accepted that advanced disease status at transplantation is a significant adverse-risk factor for post-HSCT relapse. Thus, how to improve the recurrence rate of these advanced patients after transplantation is still the main problem.

Dose intensity is a main cause for relapse. In order to improve the outcome of allo-HSCT for advanced leukemia, many scholars design the intensified conditioning or the sequential strategy of cytoreductive chemotherapy followed immediately by intensified myeloablative conditioning (MAC) regimens.With increasing dosage, the chance of relapse decreases but the incidence of acute graft-versus-host disease (GvHD) and non-relapse mortality(NRM) increase. How to well-balance NRM versus relapse is still the subject of much debate and investigation. So many centers developed reduced intensity conditioning(RIC) regimens based on the combination of alkylating agents with a purine analog and TBI, whereby the dose of TBI or the alkylating agent is usually reduced by at least 30% compared with a conventional ablative regimen. And an increased dose of alkylating agents as part of RIC may be associated with better leukemia free survival and the lower NRM.

Apart from the conditioning regimen, curative potential of allo-HSCT is largely based on immune-mediated graft-versus-leukemia(GvL)effects caused by donor T cells contained in the graft. The occurrence of GvHD is thought to be associated with a GvL effect. Since 1990, it has been known that leukemic relapses after allo-HSCT can be successfully treated by the induction of a GvL reaction. Strategies of adoptive immunotherapy such as donor lymphocyte infusion (DLI) and withdrawal of immunosuppression are proved to be able to enhance GvL effects. Many results show that the clinical benefit is limited to a minority of patients relapsed posttransplant, so new strategies such as prophylactic DLI (pDLI) before overt relapse is used in many center. But the results is varied from each centers. Liga M et reported that Patients with leukemia who received low-dose pDLI after allo-HSCT is associated with a relatively high incidence of severe GvHD. Furthermore, finding matched unrelated donors(MUD) again in a timely manner may be difficult and limit access to this treatment and the DLI process itself is more complicated.

Cyclosporine(CsA) withdrawal is generally accepted as first-line treatment in patients with relapse after allo-HSCT. In some studies, the early withdrawal of immunosuppression even in the absence of DLI, can prevent overt morphologic relapse in advanced patients.. AH Elmaagacli et al studied the immunomodulating effect of withdrawal of immunosuppression, the result showed that a probability of 10% for achieving and remaining in remission with AML 3 years after relapse posttransplant, patients with advanced CML and ALL had no chance of achieving and remaining in remission in the same time period. The best results have been seen in CML in early relapse. F Rosenow et al showed that low-tumor burden, defined by the blast count in BM aspirates, is one of the important prognostic factors for successful immune intervention. In a retrospective analysis, Sairafi et al also demonstrated that early immune intervention in case of impending relapse was more effective compared with late intervention after overt relapse. Since withdrawing immunosuppression allows for increased GvL effects, prevention may be the most feasible and effective means of managing relapse after allo-HSCT. On the basis of these results, we designed a prospective clinical study to decrease relapse risk in patients achieving CR with early reduction of immunosuppressive agents.As usual,during the first month, blood CsA levels were kept at 100-150 ng/mL in patients with sibling donors and 200-300 ng/mL in patients with a matched unrelated donors (MUD) and mismatched related donors(haplo-SCT). In the absence of GVHD, CsA was discontinued after 3-4 months when HLA-identical sibling donors were used and after 6 months when unrelated donors were used.In this clinical study,immunosuppressive agents were adjusted according to the schedule. Usually in the absence of GvHD, immunosuppressive agents were gradually reduced by 6 weeks and discontinued in three months after transplant in the advanced patients even if complete donor chimerism (CDC) achieved in matched unrelated donors(MUD) while immunosuppressive agents were gradually reduced by 2 months and discontinued in four months after transplant in the advanced patients in haploidentical SCT. If donor chimerism had not achieved CDC with no significant acute GVHD at four weeks after HSCT, immunosuppressive agents were gradually reduced. If GvHD was present during the time of immunosuppressive agents reduction, CsA was added again and tapering was done over longer periods. Immunosuppressive agents were regularly reduced by 3 months and discontinued in the 5 months without GvHD in the CR group. We used the result of chimerism as the reference. The key point in this clinicaltrial was emphasizing the early reduction of immunosuppressive agents according to the time point after transplant and the clinical symptoms. The ultimate goal of therapy is to minimize GvHD while maintaining GvL effects in order to enhance long-term disease control in the advanced patients.

ELIGIBILITY:
Inclusion Criteria: - According to the World Health Organization (WHO) classification,patients diagnosed with acute myeloid leukemia were enrolled in this study.

Performance status scores no more than 2 (ECOG criteria). Adequate organ function as defined by the following criteria: alanine transaminase （ALT）, aspartate transaminase（AST） and total serum bilirubin <2×ULN (upper limit of normal) Serum creatinine and blood urea nitrogen(BUN) <1.25×ULN. Adequate cardiac function without acute myocardial infarction, arrhythmia or atrioventricular block, heart failure, active rheumatic heart disease and cardiac dilatation(the patients has been improved after treatment of the disease and are not expected to affect transplant can include in the study).

Absence of any other contraindications of stem cell transplantation. Willingness and ability to perform HSCT. Signed and dated informed consent document indicating that the patient (or legally acceptable representative) has been informed of all pertinent aspects of the trial prior to enrollment.

Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.

Exclusion Criteria:

Presence of any condition inappropriate for HSCT. Life expectancy < 3 months because of other severe diseases. Presence of any fatal disease, including respiratory failure, heart failure, liver or kidney function failure et al.

Uncontrolled infection. Pregnancy or breastfeeding. Has enrolled in anther clinical trials Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the investigator would make the patient inappropriate for entry into this study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-01-01 (Actual); Primary Completion 2020-01-01 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
relapse free survival(RFS) | 2 years
  PFS were defined as the time from stem-cell infusion to relapse, disease progression from any cause.

SECONDARY OUTCOMES:
Progress free survival (PFS) rate | 2 years
  PFS were defined as the time from stem-cell infusion to relapse, disease progression,or death from any cause
Overall survival rate | 2 years
  OS were defined as the time from stem-cell infusion to death from any cause
Transplant related mortality | up to 2 year
  TRM were defined as death within 100 days of high-dose therapy not related to the disease,relapse or progression

CONTACTS AND LOCATIONS:
Overall Officials: xinpeng wang, doctor, Study Chair — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai First People's HOSPITAL, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Grigg AP, Szer J, Beresford J, Dodds A, Bradstock K, Durrant S, Schwarer AP, Hughes T, Herrmann R, Gibson J, Arthur C, Matthews J. Factors affecting the outcome of allogeneic bone marrow transplantation for adult patients with refractory or relapsed acute leukaemia. Br J Haematol. 1999 Nov;107(2):409-18. doi: 10.1046/j.1365-2141.1999.01713.x. PMID 10583235
- [Result] Zander AR, Dicke KA, Keating M, Vellekoop L, Culbert S, Spitzer G, Kanojia M, Jagannath S, Schell S, Hester J, et al. Allogeneic bone marrow transplantation for acute leukemia refractory to induction chemotherapy. Cancer. 1985 Sep 15;56(6):1374-9. doi: 10.1002/1097-0142(19850915)56:63.0.co;2-c. PMID 3896457
- [Result] Duval M, Klein JP, He W, Cahn JY, Cairo M, Camitta BM, Kamble R, Copelan E, de Lima M, Gupta V, Keating A, Lazarus HM, Litzow MR, Marks DI, Maziarz RT, Rizzieri DA, Schiller G, Schultz KR, Tallman MS, Weisdorf D. Hematopoietic stem-cell transplantation for acute leukemia in relapse or primary induction failure. J Clin Oncol. 2010 Aug 10;28(23):3730-8. doi: 10.1200/JCO.2010.28.8852. Epub 2010 Jul 12. PMID 20625136
- [Result] Schmid C, Schleuning M, Ledderose G, Tischer J, Kolb HJ. Sequential regimen of chemotherapy, reduced-intensity conditioning for allogeneic stem-cell transplantation, and prophylactic donor lymphocyte transfusion in high-risk acute myeloid leukemia and myelodysplastic syndrome. J Clin Oncol. 2005 Aug 20;23(24):5675-87. doi: 10.1200/JCO.2005.07.061. PMID 16110027
- [Result] Liu QF, Fan ZP, Zhang Y, Jiang ZJ, Wang CY, Xu D, Sun J, Xiao Y, Tan H. Sequential intensified conditioning and tapering of prophylactic immunosuppressants for graft-versus-host disease in allogeneic hematopoietic stem cell transplantation for refractory leukemia. Biol Blood Marrow Transplant. 2009 Nov;15(11):1376-85. doi: 10.1016/j.bbmt.2009.06.017. Epub 2009 Aug 19. PMID 19822296
- [Result] Liga M, Triantafyllou E, Tiniakou M, Lambropoulou P, Karakantza M, Zoumbos NC, Spyridonidis A. High alloreactivity of low-dose prophylactic donor lymphocyte infusion in patients with acute leukemia undergoing allogeneic hematopoietic cell transplantation with an alemtuzumab-containing conditioning regimen. Biol Blood Marrow Transplant. 2013 Jan;19(1):75-81. doi: 10.1016/j.bbmt.2012.07.021. Epub 2012 Aug 4. PMID 22871557
- [Result] Elmaagacli AH, Beelen DW, Trenn G, Schmidt O, Nahler M, Schaefer UW. Induction of a graft-versus-leukemia reaction by cyclosporin A withdrawal as immunotherapy for leukemia relapsing after allogeneic bone marrow transplantation. Bone Marrow Transplant. 1999 Apr;23(8):771-7. doi: 10.1038/sj.bmt.1701672. PMID 10231138
- [Result] Rosenow F, Berkemeier A, Krug U, Muller-Tidow C, Gerss J, Silling G, Groth C, Wieacker P, Bogdanova N, Mesters R, Buchner T, Kienast J, Berdel WE, Stelljes M. CD34(+) lineage specific donor cell chimerism for the diagnosis and treatment of impending relapse of AML or myelodysplastic syndrome after allo-SCT. Bone Marrow Transplant. 2013 Aug;48(8):1070-6. doi: 10.1038/bmt.2013.2. Epub 2013 Feb 4. PMID 23376821
- [Result] Sairafi D, Remberger M, Uhlin M, Ljungman P, Ringden O, Mattsson J. Leukemia lineage-specific chimerism analysis and molecular monitoring improve outcome of donor lymphocyte infusions. Biol Blood Marrow Transplant. 2010 Dec;16(12):1728-37. doi: 10.1016/j.bbmt.2010.06.005. Epub 2010 Jun 10. PMID 20542125
- [Derived] Yang J, Cai Y, Jiang J, Wan L, Bai H, Zhu J, Li S, Wang C, Song X. Early tapering of immunosuppressive agents after HLA-matched donor transplantation can improve the survival of patients with advanced acute myeloid leukemia. Ann Hematol. 2018 Mar;97(3):497-507. doi: 10.1007/s00277-017-3204-6. Epub 2017 Dec 18. PMID 29250743